CLINICAL TRIAL: NCT04468113
Title: Prospective, Multicenter Registry Study Evaluating the Feasibility of Ultrasound-guided Clipping of Suspicious Intramammary Lesions in Primary Breast Cancer Patients Receiving Neoadjuvant Therapy (Ultra3Detect)
Brief Title: Clip Marker Placement in Primary Lesions of Breast Cancer Patients Receiving Neoadjuvant Therapy
Acronym: Ultra3Detect
Status: Completed | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Sponsor
Other Study IDs: V2_16-04-2020
Record Dates: First submitted 2020-06-23; First posted 2020-07-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Primary Breast Cancer
Keywords: breast cancer; clip; ultrasound; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin fixed tissue from routine histopathology assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- US-guided core biopsy and clip placement: Female patients with sonographically suspicious, intramammary foci, scheduled for ultrasound-guided core biopsy and marking of the lesion with the Tumark® Vision Clip
  Interventions: Device: Tumark® Vision clip

INTERVENTIONS:
Device: Tumark® Vision clip — Suspicious intramammary lesion is marked with clip

SUMMARY:
Neoadjuvant systemic therapy (NST) is increasingly recommended for patients with early breast cancer, and the rate of patients with pathological complete remission (pCR) is increasing due to the use of modern chemotherapy regimens and targeted therapies, especially in patients with human epidermal growth factor receptor 2 positive (HER2+) breast cancer and triple negative breast cancer (TNBC). It is therefore important to mark a lesion (with e.g. clip) before the start of NST in order to safely identify and localize a clip and (former) tumor bed after completion of NST. Reliable sonographic detection of the clip would be preferred to mammography-guided detection and marking. In addition to avoiding radiation exposure by mammography and reducing time, personnel and financial expenditure, ultrasound-guided wire marking of the clip is less painful for the patient than stereotactic wire marking.

The present prospective registry study aims to evaluate how often the intramammary Tumark® Vision clip can be detected by ultrasound after completion of NST in patients with TNBC and HER2+ breast cancer and thus, in the case of pCR, how often the elaborate clipping with mammographic (stereotactic) guidance can be avoided.

DETAILED DESCRIPTION:
Breast cancer patients whose carcinomas have an aggressive tumor biology which implies the need for chemotherapy are increasingly being treated with NST. As a standard procedure, clip placement of the suspicious lesion is performed after ultrasound-guided core biopsy or mammography-guided vacuum biopsy. Clipping is necessary to enable the clear identification of the sonographically suspicious area of the breast and safe surgical removal of the remaining tumor tissue (if any) during a later surgery, even following a good response under NST. The placement of a marker (clip) is particularly important for the precise localization of the original tumor bed in patients with pCR.

There are a number of commercially available markers (clips) which are indicated for intramammary marking of a lesion and which differ in terms of shape and material. Difficulties may arise in placing the clip in the tumor or the tumor center. In addition, the clip can dislocate from the initial location and/or the clip might not be visualized during response monitoring. Evaluations of the ultrasound-visible clip made of nitinol investigated in this study showed very good results regarding marker dislocation and visibility within 7 days after inital placement.The clip, which immediately unfolds into a 3-dimensional spherical structure after insertion into the tissue, could be detected by both sonography and mammography in all 50 cases after the intervention; however, long-term data data at follow-up controls during and after NST are not available so far.

According to current German guidelines, imaging-assisted wire marking is recommended without restriction before breast conserving surgery for non-palpable lesions. The clip is considered the target lesion for wire marking, which can be done under sonographic or stereotactic control. If the clip is reliably visible on ultrasound (even in patients with pCR), the stereotactic control of wire marking can be omitted. Therefore, the ability to visualize a clip in breast ultrasonography is of great importance.

The present multicenter study aims to evaluate the sonographic detection rate of the intramammary Tumark® Vision clips after NST in clinical routine and the proportion of cases in which the clip cannot be detected, and thus the rate of mammography-guided wire markings.

ELIGIBILITY:
Inclusion Criteria:

* female patient aged ≥ 18 years
* written informed consent
* patient's consent to NST
* suspicious unilateral or bilateral intramammary foci that can be safely identified by ultrasound
* no evidence of distant metastasis (complete staging does not have to be present at inclusion)
* indication for breast conserving therapy
* no prior clip placement in the confirmed intramammary carcinoma
* patient is able to undergo NST treatment (even if the indication based on tumor biology is not yet available)
* high compliance and high number of planned relevant surgical interventions in participating study center
* patient can understand the scope of this prospective registry study

Exclusion Criteria:

* allergy to titanium and/or nickel
* pregnancy
* ipsilateral relapse (when NST: no exclusion criterion)
* prior extensive breast surgery (starting from quadrant resection)
* inflammatory breast cancer
* extramammary breast cancer
* multicentric or multifocal breast cancer
* patient is not operable
* patient is already undergoing adjuvant/neoadjuvant therapy
* inability to understand the purpose of the clinical trial or to comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with a suspicious intramammary lesion in the breast are identified as female during presentation in the clinic according to their health insurance ID card.
Study Population: Female patients with sonographically suspicious unilateral or bilateral intramammary foci, scheduled for sonography-guided core biopsy and marking of the lesion with the Tumark® Vision Clip.
Sampling Method: Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Sonographic detection rate of clip at the time of surgery after completion of NST | At the time of surgery
  Intraoperative detection rate of the clip in patients with HER2+ breast cancer or TNBC after at least 12 weeks of NST treatment

SECONDARY OUTCOMES:
Number of ultrasound-guided clip placements per patient | Immediately after placement of clip
  a) Number of lesions marked with a clip per patient and b) Number of clips per lesion
Rate of successful clip placements in the tumor center | Immediately after placement of clip
  Not successful: clip placement technically not possible or clip was placed outside the tumor (indication of the distance from the tumor center in mm)
Visibility of the device (Tumark® Vision) cannula | During placement of clip
  Visibility (very good, good, sufficient or bad) of the cannula during US-guided clip placement
Complications associated with the application of the clip | Up to 6 months after placement of clip
  e.g. hematoma, infection, dislocation, pain (in patients with or without NST)
Sonographic detection rate of clips in patients receiving NST | Immediately after placement of clip as well as after 4-8, 9-12, 13-26 weeks of NST treatment and preoperatively
  Detection rate at different time points in all patients receiving NST
Sonographic detection rate of clips in TNBC and HER2+ patients receiving NST | Immediately after clip placement as well as after 4-8, 9-12, 13-26 weeks of NST treatment and preoperatively
  Detection rate at different time points in TNBC or HER2+ breast cancer receiving NST
Sonographic detection rate of clips in all patients receiving NST and with pCR | Immediately after clip placement as well as after 4-8, 9-12,13-26 weeks of NST treatment and preoperatively
  Definition of pCR according to residual cancer burden (RCB) score
Sonographic detection rate of clips in patients not receiving NST | Immediately after clip placement and preoperatively
  Subgroup of study population not receiving NST
Intraoperative detection rate of the clip in specimen radiographs | At the time of surgery
  Detection of clip in surgical specimen from the breast subjected to radiography
Intraoperative detection rate of the clip on specimen utrasound images | At the time of surgery
  Detection of clip in surgical specimen from the breast subjected to ultrasonography
Proportion of patients requiring preoperative, mammography-guided wire marking | Preoperatively
  If ultrasound-guided wire marking is not feasible, mammography-guided wire marking is performed
Proportion of patients with mammographic verification after sonographic wire-marking | Preoperatively
  If ultrasound-guided wire marking is inconclusive
Proportion of patients with artifacts caused by clips | Up to 6 months after placement of clip
  On ultrasound and/or mammography images
Number of patients with complete pathological remission | Up to 10 weeks after surgery
  ypT0/is, ypN0 status after histological evaluation (according to Residual Cancer Burden [RCB] score) of Symmans (2007)

CONTACTS AND LOCATIONS:
Overall Officials: Sherko Kuemmel, MD, PhD, Principal Investigator — Interdisciplinary Breast Unit, Kliniken Essen-Mitte, Germany; Mattea Reinisch, MD, Study Chair — Interdisciplinary Breast Unit, Kliniken Essen-Mitte, Germany; Jörg Heil, MD, PhD, Study Chair — Department of Gynecology, Breast Center, Heidelberg University, Germany
Locations (1):
- Interdisciplinary Breast Unit, Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruland AM, Hagemann F, Reinisch M, Holtschmidt J, Kummel A, Dittmer-Grabowski C, Stoblen F, Rotthaus H, Dreesmann V, Blohmer JU, Kummel S. Using a New Marker Clip System in Breast Cancer: Tumark Vision(R) Clip - Feasibility Testing in Everyday Clinical Practice. Breast Care (Basel). 2018 Apr;13(2):116-120. doi: 10.1159/000486388. Epub 2018 Mar 9. PMID 29887788
- [Background] Hurvitz SA, Martin M, Symmans WF, Jung KH, Huang CS, Thompson AM, Harbeck N, Valero V, Stroyakovskiy D, Wildiers H, Campone M, Boileau JF, Beckmann MW, Afenjar K, Fresco R, Helms HJ, Xu J, Lin YG, Sparano J, Slamon D. Neoadjuvant trastuzumab, pertuzumab, and chemotherapy versus trastuzumab emtansine plus pertuzumab in patients with HER2-positive breast cancer (KRISTINE): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2018 Jan;19(1):115-126. doi: 10.1016/S1470-2045(17)30716-7. Epub 2017 Nov 23. PMID 29175149
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Background] Shah AD, Mehta AK, Talati N, Brem R, Margolies LR. Breast tissue markers: Why? What's out there? How do I choose? Clin Imaging. 2018 Nov-Dec;52:123-136. doi: 10.1016/j.clinimag.2018.07.003. Epub 2018 Jul 6. PMID 30059952